CLINICAL TRIAL: NCT05535010
Title: The Effect of the Presence of Active Trigger Points in the Muscles Innervated by the Affected Nerve Roots on the Treatment Results of Transforaminal Epidural Steroid Injection in Patients With Lumbar Radiculopathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04.03.2022.473
Record Dates: First submitted 2022-07-01; First posted 2022-09-10 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-07

CONDITIONS: Trigger Point Pain, Myofascial; Lumbar Radiculopathy
Keywords: Trigger point; Myofascial; Lumbar radiculopathy; Transforaminal epidural steroid injection
MeSH Terms: conditions — Myofascial Pain Syndromes; Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Those with active trigger points before TFESI (Experimental): Transforaminal epidural steroid injection
  Interventions: Procedure: Transforaminal epidural steroid injection(TFESI)
- Those who do not have an active trigger point before TFESI (Active Comparator): Transforaminal epidural steroid injection
  Interventions: Procedure: Transforaminal epidural steroid injection(TFESI)

INTERVENTIONS:
Procedure: Transforaminal epidural steroid injection(TFESI) — TFESI procedure will be applied again in the 3rd week and 3rd month for the patients whose NRS score decreased by less than 50 percent after the first procedure.

SUMMARY:
The association between lumbosacral radiculopathy and the ipsilateral gluteal trigger point has been demonstrated in 74% of previous studies in patients with chronic low back pain. It has also been found to be associated with lumbosacral radiculopathy, central sensitization and myofascial pain in previous studies.

From these data, it can be hypothesized that the presence of a myofascial trigger point in the relevant muscle segment may alter the efficacy of the transforaminal epidural steroid injection (TFESI) procedure used in the treatment of lumbosacral radiculopathy. We could not find any study on this subject in the literature. Although the most accurate level for the TFESI procedure is determined according to the patient's examination and imaging findings, patients may not benefit from the procedure sufficiently due to the trigger points on the same side as the radicular pain before the procedure. Another hypothesis is that active trigger points will transform into latent or normal tissue after the TFESI procedure and patients will benefit significantly. This assumption will provide insight into the possible underlying mechanism in some patients who do not benefit from the TFESI procedure. If the active trigger points become latent or there is a significant change in the pressure pain threshold after the TFESI procedure, the formation mechanism of the trigger points will be understood.

TFESI is one of the procedures routinely applied to patients diagnosed with lumbosacral radiculopathy in investigator's clinic. Among the patients who are planned to undergo TFESI procedure, those who are suitable for our study will be selected. Data such as demographic characteristics, height, weight, which leg the pain is reflected in, additional diseases, medications, the stage of the disc herniation, pressure on which nerve root, presence and number of active trigger points, muscles will be recorded before the procedure. Numerical Rating Scale (NRS), Short Form-12, Central Sensitivity Inventory (CSI), Doulour Neuropathic 4 (DN4), 6-point Likert Scale, Jenkins Sleep Scale, Istanbul Low Back Pain Disability Index, Pressure Pain Threshold (active trigger points will be evaluated with an algometer) will be applied to the patients before the procedure. The patients will be evaluated for the presence of active trigger points before the procedure and the patients will be divided into 2 groups as those with active trigger points and those without. The same procedure will be applied to both groups as planned before inclusion of the patients in the study, in the same way as the patients ineligible for the study. Patients will be re-evaluated with the scales and methods mentioned above at the 3rd week, 3rd and 6th months after the first procedure. TFESI procedure will be performed again in the 3rd week and 3rd month for the patients whose NRS values decrease less than 50 percent after the previous procedure.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain for at least 3 months due to lumbosacral radiculopathy
* Root compression due to paracentral disc herniation at L4-L5 or L5-S1 levels in accordance with the patient's complaint and clinical findings in lumbar MRI imaging
* Being unresponsive to conservative treatment
* Volunteering to participate in the study and signing a consent form

Exclusion Criteria:

* History of surgery on the lumbar region/interventional procedure in the last 6 months
* Presence of additional musculoskeletal disease (such as lateral epicondylitis, tendinitis)
* Disease that may change the anatomical or physiological structure of the relevant regions (such as rheumatoid arthritis, osteoporosis)
* Presence of coagulopathy
* Presence of lumbar spinal stenosis
* Having a diagnosis of fibromyalgia
* Being pregnant or breastfeeding
* History of allergy to the injectables to be administered
* Having a diagnosis of mental, psychiatric or neurological disease that may complicate the application of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-04-02 (Estimated); Study Completion 2023-04-02 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | 3 months
  NRS is a scale in which the patient gives points between "0" and "10" for the low back and leg pain felt by the patient, "0" = No pain, "10" = The most severe, unbearable pain

SECONDARY OUTCOMES:
Short Form-12 | 3 weeks, 3 and 6 months
  SF-12 is a scale that evaluates the patient's quality of life
Central Sensitization Inventory (CSI) | 3 weeks, 3 and 6 months
  The central sensitization scale is a two-part scale that evaluates the patient's neuropathic complaints and records the associated diagnosis, if any
Doulour Neuropathic 4 (DN4) | 3 weeks, 3 and 6 months
  DN4 is a scale that evaluates the patient's neuropathic symptoms with 4 questions.
6-point Likert Scale | 3 weeks, 3 and 6 months
  A 6-point Likert scale is based on patient expression ''1 ''= I am much worse, ''2'' = I am slightly worse, ''3''= I am the same, ''4''= I am slightly better, '' 5''= I am much better, ''6''= I am completely better
Jenkins Sleep Scale | 3 weeks, 3 and 6 months
  The Jenkins Sleep Scale is a 4-item scale that evaluates sleep.
Pressure Pain Threshold | 3 weeks, 3 and 6 months
  Pressure pain threshold is a value measured with an algometer, applied to the skin from an area of 1 cm2, and recording the pressure value at which the person feels pain with increasing pressure.
Istanbul Low Back Pain Disability Index | 3 weeks, 3 and 6 months
  Istanbul Low Back Pain Disability Index, on the other hand, is a scale that evaluates the effect of low back pain on the daily life of a person with 18 questions.
Number of trigger points | 3 weeks, 3 and 6 months
  Number of trigger points in muscles innervated by L5 and S1 roots

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No